CLINICAL TRIAL: NCT06238921
Title: Phase I/II Study of Stereotactic Radiation and Sacituzumab Govitecan With Zimberelimab in the Management of Metastatic Triple Negative Breast Cancer With Brain Metastases (TARGET-TNBC)
Brief Title: Sacituzumab Govitecan and Zimberelimab w/SRS in the Management of Metastatic Triple Negative Breast Cancer With Brain Metastases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21676
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Radiosurgery; zimberelimab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SG + Zimberelimab with SRS (Experimental): Treatment will be initiated with SRS followed 1 week later by SG on days 1 and 8 (10mg/kg) with zimberelimab on day 1 (360 mg IV) repeated every 3 weeks follow-up imaging response assessments will be conducted at q9 week intervals.
  Interventions: Radiation: Stereotactic Radiation; Drug: Zimberelimab; Drug: Sacituzumab govitecan

INTERVENTIONS:
Radiation: Stereotactic Radiation — Stereotactic Radiation to intact brain metastases or post-operative cavity.
Drug: Zimberelimab — One week +/- 4 days following receipt of SRS, zimberelimab 360 mg IV will be administered. This will be followed by zimberelimab 360 mg IV every 3 weeks.
Drug: Sacituzumab govitecan — SG will be administered on days 1 and 8 (10 mg/kg) of 21 day treatment cycles. This will be one week +/- 4 days following receipt of SRS for the first dose.
  Other Names: Trodelvy

SUMMARY:
This is a Phase I/II Study to determine the safety and efficacy of Sacituzumab Govitecan and Zimberelimab with stereotactic radiation (SRS) in participants with metastatic triple negative breast cancer with brain metastases, compared to treatment with Sacituzumab Govitecan alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated Informed Consent Form (ICF).
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Age ≥ 18.
* Triple negative breast cancer; to fulfill the requirement of triple negative disease, a breast cancer must express (≤ 10%), by immunohistochemistry (IHC), of the hormone receptors (estrogen receptor [ER] and progesterone receptor [PR]).
* Breast cancer as documented by extracranial tumor biopsy with brain metastases documented from MRI brain imaging or intracranial surgical pathology.
* Eligible for Stereotactic radiosurgery (SRS) to brain metastases or to the post-operative bed.
* Measurable brain disease per RANO-BM criteria1 that can be measured in at least one dimension as ≥ 0.5 cm for both intact brain metastases and post-operative cavities.
* Maximum diameter of the largest intact brain metastases ≤ 4 cm.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Symptomatic patients having undergone surgery or on stable doses of steroids ≤ 8 mg/day dexamethasone will be enrolled.
* Prior treatment with taxane based chemotherapy with anthracyclines.
* Individuals with prior SRS/fractioned stereotactic radiotherapy (FSRT) treatment will be allowed if active measurable disease has not previously been treated with radiation therapy.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the administration of each dose of study agent.
* Male and female patients of childbearing potential who engage in heterosexual intercourse must agree to use specified method(s) of contraception.

Exclusion Criteria:

* Presence of leptomeningeal disease.
* Women who are pregnant or breastfeeding.
* Known history of HIV-1 or 2 with detectable viral load.
* Active, known, or suspected autoimmune disease. Patients with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded. Exceptions are patients with type I diabetes mellitus, hypothyroidism only requiring thyroid replacement therapy, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Met any of the following criteria for cardiac disease:

  1. Myocardial infarction or unstable angina pectoris within 6 months of enrollment
  2. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation
  3. New York Heart Association (NYHA) Class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
* Any patient requiring supplemental oxygen therapy.
* Have an active serious infection requiring antibiotics.
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
* Patients with prior history of non-breast cancer malignancies are excluded except in the case of adequately treated basal cell cancer, squamous cell skin cancer, chronic lymphocytic leukemia, or other cancers in remission not receiving active therapy for ≥ 2 years.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or that would interfere with the interpretation of safety results.
* Major surgery or significant traumatic injury that has not been recovered from by 14 days before the initiation of study drug.
* Have had a prior anticancer biologic agent within 4 weeks prior to enrollment or have had prior chemotherapy, targeted small molecule therapy within 2 weeks prior to enrollment and have not recovered.
* Have previously received topoisomerase 1 inhibitors in the setting of brain metastases.
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.
* Have active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.
* History of allergy or hypersensitivity to any of the study drugs or study drug components.
* Prisoners or individuals who are involuntarily incarcerated.
* Individuals who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Phase I: Neurologic Toxicity | Up to 9 Weeks
  Neurologic Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5). A Neurologic Toxicity will be defined as any Grade 3 or higher toxicity that occurs during the Dose Limiting Toxicity evaluation period. Toxicity that is clearly and directly related to the primary disease or to another etiology is excluded from this definition.
  * Symptomatic radionecrosis, defined by surgical pathology or multidisciplinary evaluation.
  * Grade ≥ 3 headaches
  * Grade ≥ 3 memory impairment
  * New onset grade ≥ 3 seizures
Phase II: Progression Free Survival (PFS) | Up to 12 Months
  Evaluate the PFS of SG and zimberelimab with SRS among patients with metastatic triple negative breast cancer.
  PFS is time from the date of start of treatment to the investigator-determined date of progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Phase II: Intracranial Progression Free Survival (PFS) | Up to 12 Months
  Time from the date of start of treatment to the investigator-determined date of progression (determined by Response Assessment in Neuro-Oncology (RANO)) or death due to any cause, whichever occurs first.
  Progression is measured by a ≥ 20% increase in sum longest distance relative to nadir in target lesions and unequivocal or progressive disease in non-target lesions.
Phase II: Extracranial Progression Free Survival (PFS) | Up to 33 Months
  PFS will be measured from the date of start of treatment to the investigator-determined date of progression (determined by Immune-related Response Evaluation Criterial in Solid Tumors (irRECIST)) or death due to any cause, whichever occurs first.
  Progression is defined as ≥ 20% increase in tumor burden.
Phase II: Overall Survival (OS) | Up to 33 Months
  OS will be measured from the date of start of treatment to death.
Phase II: Local Brain Control | Up to 33 Months
  Number of participants with Local Brain Control will be determined from irradiated lesions according to RANO criteria.
Phase II: Distant Brain Control | Up to 33 months
  Number of participants with Distant Brain Control will be determined by the development of new lesions outside the irradiated area.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No